CLINICAL TRIAL: NCT03401723
Title: A Validation Study of the 3D-CoPS and 3D-CoRS and Its Relationship With an International Acknowledged Assessment Tool (ETS) in Simulated Colonoscopy
Brief Title: A Validation Study of a Computerized Movement Analysis of the Colonoscope in Simulated Colonoscopy
Acronym: 3D-CoPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Technical University of Denmark (Other)
Responsible Party: Principal Investigator, Andreas Slot Vilmann, MD. Andreas Slot Vilmann, Rigshospitalet, Denmark
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 3D-CoPS and 3D-CoRS
Record Dates: First submitted 2017-12-22; First posted 2018-01-17 (Actual); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Education
Keywords: Validation study; Simulation; Endoscopy

STUDY DESIGN:
Masking Description: This is a vialidation study of a computerized analysis of the colonoscope movements during a simulated procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Novices (Other): Any physician who has no experience of endoscopies or has done no more than 50 colonoscopies.
  Each subject included are to perform on the Endoscopy Training System (ETS) during which data for 3D-Colonoscopy Progression Score and 3D-Colonoscopy Retraction Score is gathered.
  Interventions: Other: 3D-Colonoscopy Progression Score; Other: Endoscopy Training System; Other: 3D-Colonoscopy Retraction Score
- Experienced (Other): Includes any physician who have succeeded more than 140 colonoscopies. Professional backgrounds include surgeons and gastroenterologists.
  Each subject included are to perform on the ETS during which data for 3D-Colonoscopy Progression Score and 3D-Colonoscopy Retraction Score is gathered.
  Interventions: Other: 3D-Colonoscopy Progression Score; Other: Endoscopy Training System; Other: 3D-Colonoscopy Retraction Score

INTERVENTIONS:
Other: 3D-Colonoscopy Progression Score — 3D-Colonoscopy Progression Score is a computerized analysis of the movement of the colonoscope based on data from coils within the colonoscope.
  Other Names: 3D-CoPS
Other: Endoscopy Training System — The Endoscopy Training System is based on the Colonoscopy Training Model platform and includes four different performance metrics and a scoring system.
  1. Scope Manipulation - The use of torque and tip deflection to move a shape in the colon
  2. Tool Targeting - 10 targets located around the colon must be found. With a biopsy forceps, each target has to been touched.
  3. Loop Management - The management of a standard alfa-loop.
  4. Mucosal Inspection - Randomly placed polyps inside the rubber colon have to be found during withdrawal.
  Other Names: ETS
Other: 3D-Colonoscopy Retraction Score — 3D-Colonoscopy Retraction Score is a computerized analysis of the movement of the colonoscope based on data from coils within the colonoscope.
  Other Names: 3D-CoRS

SUMMARY:
A cross validation study comparing an international acknowledged assessment tool "Endoscopy Training System" (ETS) and movement analysis of the colonoscope based on raw data from coils within the scope.

24 physicians are recruited and divided based on experience (novices and experienced). All participants are to perform twice on the ETS that is based on four tasks; Scope manipulation, tool targeting, loop management and mucosal inspection. The movement of the colonoscope will be gathered during the tasks and correlated to the scores of the ETS.

DETAILED DESCRIPTION:
24 physicians are recruited on a voluntarily basis, and will be divided into two groups, based on experience;

1. 12 Novices (0-50 colonoscopies)
2. 12 Experienced (> 140 colonoscopies). The groups are to perform twice on the Endoscopy Training System that is based on four tasks; Scope manipulation, tool targeting, loop management and mucosal inspection. Data for 3D-Colonoscopy Retraction Score (3D-CoRS) will be gathered during the task of mucosal inspection and data for 3D-Colonoscopy Progression Score (3D-CoPS) are collected during loop management.

Novice group:

Any physician who has no experience of endoscopies or has done no more than 50 colonoscopies.

Experienced group:

Includes any physician who have succeeded more than 140 colonoscopies. Professional backgrounds include surgeons and gastroenterologists.

Demographic data will gathered from all three groups as follows:

* Age
* Sex
* Speciality
* Total number of colonoscopies
* Total number of colonoscopies the last year
* Time since graduation
* Experience in simulated endoscopy/colonoscopy The Endoscopy Training System is a simulation system and an assessment tool and includes five different performance metrics and a scoring system. The system is used in combination with an Olympus colonoscope (Olympus Medical Systems Corp. Tokyo, Japan).

Performance metrics:

1. Scope Manipulation (SM) - The use of torque and tip deflection to move a shape in the colon to the 6 o´clock position and align the same shape within an outline placed upon the monitor screen. Before continuing to the next shape, alignment must be held for 5 seconds.
2. Tool Targeting (TT) - 10 targets located around the colon must be found. With a biopsy forceps, each target has to been touched for at least 5 seconds before moving to the next target.
3. Loop Management (LM) - The management of a standard alfa-loop. If during insertion from anus until cecum a loop is formed, it must be first recognised and then unlooped successfully to continue advancing the colonoscope.

   The Colonoscopy Training Model begin in the left lateral position, but on request, the model can be repositioned in the supine, prone, or right lateral decubitus position. On request, abdominal pressure can be provided when directed by the participant.
4. Mucosal Inspection (MI) - Randomly placed polyps inside the rubber colon have to be found during withdrawal, requiring inspection and retroflexion in the rectum.
5. Retroflexion (RF) - 5 targets located around the anus must be found. With a biopsy forcep, each target has to been touched while the colonoscope is retroflexed in the rectum and touched for at least 5 seconds before moving to the next target.

The 3D-Colonoscopy Progression Score (3D-CoPS) and the 3D-Colonoscopy Retraction Score (3D-CoRS) are movement analysis. Electromagnetic coils are built in along the length of the Olympus colonoscopes. They generate a pulsed low-intensity magnetic field that is picked up a receiver coil. The data-points for each coil are inserted into an algorithm for movement analyzing. This analysis is done as a change between the tip of the scope, and the next tracked magnetic coil. The result is a relative movement of the colonoscope in relation to the previous position, and how much the movement is deflected according to the direction the tip points in. This movement analysis is used for distinction between the progression- and retraction phase, and as the basis for the 3D-CoPS and 3D-CoRS analysis, which is essential, such that the 3D-CoRS measurements is performed during withdrawal of the colonoscope.

ELIGIBILITY:
Inclusion Criteria:

* Physicians

Exclusion Criteria:

* Non physicians

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-03-21 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
3D-Colonoscopy Progression Score | 3 months
  The score is based on a movement analysis of the colonoscope from anus until max insertion(cecum). It is scaled from 0-1000 .A score of zero equals an incomplete procedure and a score of 1 is a very poor score but the cecum was reached. Increasing score represents better technical performance with a maximum score of 1000.
3D-Colonoscopy Retraction Score | 3 months
  The score is based on a movement analysis of the colonoscope from cecum to the anus. It is scaled from 0-1000. A score of zero equals a very poor score, Increasing score represents better technical performance with a maximum score of 1000.

SECONDARY OUTCOMES:
Relationship to other variables | 3 months
  Scores from the ETS, 3D-CoPS and 3D-CoRS will be correlated.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Konge, Prof, Study Director — CAMES-Rigshospitalet
Locations (1):
- Copenhagen Acedemy of Medical Education and Simulation, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ritter EM, Cox TC, Trinca KD, Pearl JP. Simulated Colonoscopy Objective Performance Evaluation (SCOPE): a non-computer-based tool for assessment of endoscopic skills. Surg Endosc. 2013 Nov;27(11):4073-80. doi: 10.1007/s00464-013-3063-8. Epub 2013 Jul 17. PMID 23860607
- [Background] Trinca KD, Cox TC, Pearl JP, Ritter EM. Validity evidence for the Simulated Colonoscopy Objective Performance Evaluation scoring system. Am J Surg. 2014 Feb;207(2):218-25. doi: 10.1016/j.amjsurg.2013.08.026. Epub 2013 Oct 23. PMID 24246259